CLINICAL TRIAL: NCT04806477
Title: Randomized Trial of Diagnostic Accuracy of Medical Evaluation by Telemedicine Compared to Face-to-face Medical Evaluation in an Emergency Care Unit in Immunocompetent Adult Patients With Symptoms Suggestive of Acute Airway Infection
Brief Title: Diagnostic Accuracy Comparison Between Telemedicine and Face-to-face Consultations in Respiratory Infection Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 34172720400000071
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Tract Infections
Keywords: Telemedicine; Respiratory Tract Infections; Emergency Medical Services; Referral and Consultation; COVID-19
MeSH Terms: conditions — Respiratory Tract Infections; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult patients with respiratory tract symptom - telemedicine before face-to-face evaluation (Active Comparator): We included adults (≥18 years of age) who had at least one acute symptom compatible with Respiratory Tract Infection (sore throat, nasal obstruction, coryza, new or growing cough, sputum, hoarseness, dyspnea) with or without symptoms related to the infection (fever ≥ 38oC, chills, sweating, myalgia) who have undergone telemedicine consultation before face-to-face evaluation
  Interventions: Other: Telemedicine Consultation; Other: Face-to-face Consultation
- Adult patients with respiratory tract symptom - only face-to-face evaluation (Active Comparator): We included adults (≥18 years of age) who had at least one acute symptom compatible with Respiratory Tract Infection (sore throat, nasal obstruction, coryza, new or growing cough, sputum, hoarseness, dyspnea) with or without symptoms related to the infection (fever ≥ 38oC, chills, sweating, myalgia) who have undergone only face-to-face evaluation
  Interventions: Other: Face-to-face Consultation

INTERVENTIONS:
Other: Telemedicine Consultation — Brief telemedicine consultation, blinded to subsequent face-to-face evaluation.
  Arms: Adult patients with respiratory tract symptom - telemedicine before face-to-face evaluation
Other: Face-to-face Consultation — Direct face-to-face evaluation (without telemedicine consultation before).

SUMMARY:
This is a randomized study that sought to analyze the diagnostic accuracy of the telemedicine consultation of patients suspected of respiratory tract infections during COVID-19 pandemic in comparison with the face-to-face evaluation at the emergency department.

DETAILED DESCRIPTION:
Unicentric, prospective and randomized study performed between September and November 2020 with adult patients who sought care at emergency department. The inclusion criterion was the exhibition of any tract respiratory symptom. Patients older than 65 years, with chronic heart or lung diseases or immunosuppressed were excluded. Eligible patients were randomized 1:1 for a brief telemedicine consultation, blinded to subsequent face-to-face evaluation or direct face-to-face evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one acute symptom compatible with RTI (sore throat, nasal obstruction, coryza, new or growing cough, sputum, hoarseness, dyspnea) in presence or absence of symptoms related to the infection (fever ≥ 38oC, chills, sweating, myalgia) that motivated spontaneously face-to-face evaluation at the ED.

Exclusion Criteria:

* Patients with diagnosis of chronic respiratory diseases (chronic obstructive pulmonary disease, asthma and interstitial lung disease)
* Patients with previous diagnosis of congestive heart failure,
* Patients with HIV / AIDS
* Patients with active cancer
* Patients with type I diabetes mellitus
* Patients in use of any immunosuppressant
* Patients with chronic cough
* Patiets that referral to emergency room after nursing triage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Number of final evaluation ICD 10-code diagnosis. | up to 10 months
  All institutional Emergency Department or Telemedicine assessments involve filling out the final diagnosis on an International Classification of Diseases (ICD-10)-code basis in the electronic medical record before discharge to home or admission. For aggregation of most prevalent RTI with similar pathophysiologic characteristics, three diagnostic groups were defined, based on ICD 10 codes: RTI, including COVID-19 (B34.2, B34.9, B97.2, J00, J04, J06, J11, J20, J30, J39, U07.1); PT - Acute Pharyngotonsillitis (J02-J03.9) and AS - Acute Sinusitis (J01-J01.9).

SECONDARY OUTCOMES:
Time of medical care | up to 10 months
  Comparison of time (minutes) of medical care between telemedicine and face-to-face consultation.
Rate of indication for complementary exams | up to 10 months
  Comparison of rate (percentage) of indication for complementary exams between telemedicine and face-to-face consultation.
Type of requested exams | up to 10 months
  Comparison of type of requested exams (porcentage) between telemedicine and face-to-face consultation.
Type of Medical prescription | up to 10 months
  Comparison of type of medical prescription after completion of the service between telemedicine and face-to-face consultation
Type of proposed destination after completion of the service | up to 10 months
  Comparison of proposed destination (percentage of discharge or hospitalization) after completion of the service between telemedicine and face-to-face consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo HS Cordioli, MD, Study Director — Telemedicine Department, Hospital Israelita Albert Einstein, Sao Paulo, Brazil
Locations (1):
- Hospital Israelita Abert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Accorsi TAD, Moreira FT, Pedrotti CHS, Amicis K, Correia RFV, Morbeck RA, Medeiros FF, Souza JL Jr, Cordioli E. Telemedicine diagnosis of acute respiratory tract infection patients is not inferior to face-to-face consultation: a randomized trial. Einstein (Sao Paulo). 2022 May 27;20:eAO6800. doi: 10.31744/einstein_journal/2022AO6800. eCollection 2022. PMID 35649057